CLINICAL TRIAL: NCT01814969
Title: Preoperative Hyperfractionated Radiotherapy Versus Combined Radiochemotherapy for Patients With Locally Advanced Rectal Cancer: a Phase III Randomized Trial.
Brief Title: Preoperative Hyperfractionated Radiotherapy or Radiochemotherapy in Locally Advanced Rectal Cancer.
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Maria Sklodowska-Curie National Research Institute of Oncology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PHRT-COI-01
Record Dates: First submitted 2013-03-18; First posted 2013-03-20 (Estimated); Last update posted 2015-05-05 (Estimated); Status verified 2015-05

CONDITIONS: Rectal Cancer
Keywords: Rectal neoplasm; Preoperative hyperfractionated radiotherapy; Preoperative hyperfractionated radiochemotherapy
MeSH Terms: conditions — Rectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Hyperfractionated Radiochemotherapy (Experimental): radiotherapy in rectal tumor area due to the placing of pelvic nodal groups to a total dose of 42 Gy, 1.5 Gy d fx 2 times a day; (gap between the factions min. 6-8h) - duration of treatment 2.5 weeks with simultaneous two cycles of chemotherapy according to the scheme: 5FU-325mg/m2 (bolus) on 1-3 and 16-18 (last 3 days of radiotherapy).
  Surgical resection has to be done within 14 days or 5-6 weeks after the completion of hyperfractionated radiochemotherapy (HRTCT).
  Interventions: Radiation: Hyperfractionated Radiochemotherapy
- Hyperfractionated Radiotherapy (Active Comparator): radiotherapy in rectal tumor area due to the placing of pelvic nodal groups to a total dose of 42 Gy, 1.5 Gy d fx 2 times a day; (gap between the factions min. 6-8h) - duration of treatment 2.5 weeks.
  Surgical resection has to be done within 14 days or 5-6 weeks after the completion of hyperfractionated radiotherapy (HRT).
  Interventions: Radiation: Hyperfractionated Radiotherapy

INTERVENTIONS:
Radiation: Hyperfractionated Radiochemotherapy — 28 x 1.5Gy 2 times a day; gap between the fractions min. 6-8h - duration of treatment 2.5 weeks + simultaneous bolus 5-Fluorouracil (the each cycle consisted of 5-fluorouracil 325 mg/m2 per day) on 1-3 and 16-18 (last 3 days of radiotherapy).
  Other Names: Hyperfractionated Radiochemotherapy (HRTCT)
  Arms: Hyperfractionated Radiochemotherapy
Radiation: Hyperfractionated Radiotherapy — 28 x 1.5Gy 2 times a day; gap between the factions min. 6-8h - duration of treatment 2.5 weeks
  Other Names: Hyperfractionated Radiotherapy (HRT)
  Arms: Hyperfractionated Radiotherapy

SUMMARY:
Clinical objective of the study is to compare the rates of pathologic response, acute toxicity and sphincter preservation with two schedules of preoperative regiment in patients with locally advanced rectal cancer.

DETAILED DESCRIPTION:
Overview of randomized trials conducted in patients with advanced colorectal cancer with the use of preoperative radiotherapy or radiochemotherapy clearly shows the superiority of combined therapy over surgery alone. In these studies documented a significant reduction in tumor mass as a result of preoperative radiotherapy or radiochemotherapy theoretically increases the chance of performing operations with sphincters preservation, even in cases originally eligible for abdomino - perineal resection. There is the question whether the combination of preoperative hyperfractionated radiotherapy and concurrent chemotherapy may cause the further improvement of treatment outcome in patients with locally advanced rectal cancer. Published in 2012 by Gerard et al. meta-analysis of randomized trials dedicated to the treatment of patients with advanced colorectal cancer, confirms a higher percentage of sphincters preservation in patients operated after more than 5-week interval between neoadjuvant therapy and surgery.

Analysis of these issues will be taken in the current study. Comparison of the two treatment regimens as preoperative phase III study with stratification for time interval between the end of radiotherapy or radiochemotherapy and surgery may show differences that have not been seen in previously published data.

ELIGIBILITY:
Inclusion Criteria:

1. Karnofsky Index 80% or better (Zubrod 0-1)
2. Histological proved diagnosis of rectal cancer (adeno- or mucinous carcinoma)
3. Primary rectal cancer:

   3.1. Maximum 12 cm above dentate line (upper limit) 3.2. Staged T2N+ or T3N0 or T3N+ (by endorectal ultrasound or Computed Tomography [CT]/Magnetic Resonance Imaging [MRI] scan)
4. No evidence of metastatic disease as determined by chest X-ray and abdominal ultrasound (or CT-scan of chest and abdomen or other investigations such as Positron Emission Tomography [PET] scan or biopsy if required)
5. Adequate bone marrow function with platelets more than 100 × 10^9/l and neutrophils more than 2.0 × 10^9/l
6. Creatinine clearance more than 50 ml/min
7. Serum bilirubin less than 2.0 × Upper Limit of institutional Normal range (ULN)
8. Written informed consent is obtained prior to commencement of trial treatment (confirmed the signature on the consent form for the proposed project and the standard medical consent form for radiotherapy within the abdominal cavity).

Exclusion Criteria:

1. Rectal cancer other than adeno- or mucinous carcinoma
2. Previous or concurrent malignancies, with the exception of adequately treated basal cell carcinoma of the skin
3. Patients with locally advanced inoperable disease, such as T4-tumour
4. Presence of metastatic disease or recurrent rectal tumour
5. Any previous chemotherapy or radiotherapy, and any investigational treatment for rectal cancer
6. Concurrent uncontrolled medical conditions
7. Pregnancy or breast feeding
8. Clinically significant (i.e. active) cardiac disease (e.g. congestive heart failure, symptomatic coronary artery disease) or myocardial infarction within the last six months
9. Evidence of hereditary colorectal cancer (Hereditary Non-Polyposis Colorectal Cancer [HNPCC] and Familial Adenomatous Polyposis [FAP])
10. Medical or psychiatric conditions that compromise the patient's ability to give informed consent
11. No agreement for randomisation

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 260 (Estimated)
Dates: Start 2014-03; Primary Completion 2016-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
• The rate of patients with downstaging after radiotherapy or radiochemotherapy to pathological response or disease with negative margins | Surrogate endpoint available immediatly after surgery

SECONDARY OUTCOMES:
The rate of local failures | 3 years
Progression-free long-term survival | 3 years
The rate of distant metastases | 3 years
Overall long-term survival | 3 years
The rate of late toxicity according to the RTOG/EORTC scale | 3 years
The rate of postoperative complications | 3 months
The rate of early toxicity of neoadjuvant treatment according to the NCI CTCAE (version 4.0) | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Rafal Suwinski, MD, Principal Investigator — Maria Sklodowska-Curie Memorial Cancer Center and Institute of Oncology, Gliwice Branch, Gliwice, Poland
Locations (1):
- Maria Sklodowska-Curie Memorial Cancer Center and Institute of Oncology Gliwice Branch, Gliwice, Wybrzeze AK 15, Poland

REFERENCES:
- [Background] Suwinski R, Wzietek I, Tarnawski R, Namysl-Kaletka A, Kryj M, Chmielarz A, Wydmanski J. Moderately low alpha/beta ratio for rectal cancer may best explain the outcome of three fractionation schedules of preoperative radiotherapy. Int J Radiat Oncol Biol Phys. 2007 Nov 1;69(3):793-9. doi: 10.1016/j.ijrobp.2007.03.046. Epub 2007 May 17. PMID 17499451
- [Background] Suwinski R, Wydmanski J, Pawelczyk I, Starzewski J. A pilot study of accelerated preoperative hyperfractionated pelvic irradiation with or without low-dose preoperative prophylactic liver irradiation in patients with locally advanced rectal cancer. Radiother Oncol. 2006 Jul;80(1):27-32. doi: 10.1016/j.radonc.2006.05.001. Epub 2006 May 26. PMID 16730087
- [Background] Gerard JP, Rostom Y, Gal J, Benchimol D, Ortholan C, Aschele C, Levi JM. Can we increase the chance of sphincter saving surgery in rectal cancer with neoadjuvant treatments: lessons from a systematic review of recent randomized trials. Crit Rev Oncol Hematol. 2012 Jan;81(1):21-8. doi: 10.1016/j.critrevonc.2011.02.001. Epub 2011 Mar 5. PMID 21377377
- [Derived] Idasiak A, Galwas-Kliber K, Rajczykowski M, Debosz-Suwinska I, Zeman M, Stobiecka E, Mrochem-Kwarciak J, Suwinski R. Tumor regression grading after preoperative hyperfractionated radiotherapy/chemoradiotherapy for locally advanced rectal cancers: interim analysis of phase III clinical study. Neoplasma. 2021 May;68(3):631-637. doi: 10.4149/neo_2021_201217N1366. Epub 2021 Feb 24. PMID 33618522
- [Derived] Idasiak A, Galwas-Kliber K, Behrendt K, Wzietek I, Kryj M, Stobiecka E, Chmielik E, Suwinski R. Pre-operative hyperfractionated concurrent radiochemotherapy for locally advanced rectal cancers: a phase II clinical study. Br J Radiol. 2017 Jun;90(1074):20160731. doi: 10.1259/bjr.20160731. Epub 2017 May 23. PMID 28466686